CLINICAL TRIAL: NCT01588236
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Phase 2 Study to Further Assess the Efficacy, Safety and Dose Response of KYG0395 in the Treatment of Primary Dysmenorrhea
Brief Title: Effect of KYG0395 on Primary Dysmenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GF-2011-001
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- high dose KYG0395 (Experimental): Patients received high dose KYG0395 capsule (tid)
  Interventions: Drug: high dose KYG0395
- lower dose KYG0395 (Experimental): Patients received lower dose KYG0395 capsule (bid)
  Interventions: Drug: lower dose KYG0395
- placebo (Placebo Comparator): Patients received placebo (tid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: high dose KYG0395 — 3 KYG0395 capsules tid (morning, midday, and evening)
  Other Names: KYG0395 high dose
  Arms: high dose KYG0395
Drug: lower dose KYG0395 — 3 KYG0395 capsules 2 times a day (bid) (morning and evening) plus 3 capsules of placebo (midday)
  Other Names: KYG0395 low dose
  Arms: lower dose KYG0395
Drug: Placebo — 3 capsules of placebo tid (morning, midday, and evening)
  Other Names: Placebo oral capsule
  Arms: placebo

SUMMARY:
The purpose of this study is to further assess the efficacy, safety and dose-response of KYG0395 in the treatment of primary dysmenorrhea.

DETAILED DESCRIPTION:
Compare the effect and safety of the investigational drug and placebo on dysmenorrhea in adult otherwise healthy women.

ELIGIBILITY:
Inclusion Criteria:

1. Reviewed and signed the ICF.
2. Female between the ages of 18 and 35 (inclusive) at the time of signing the ICF.
3. Otherwise healthy female subjects with primary dysmenorrhea for at least 3 consecutive menstrual cycles prior to the study (prior to the start of the baseline cycles) and with VAS score >70 for the maximum dysmenorrheic pain or VAS score >40 for the average daily dysmenorrheic pain of the last menstrual cycle.
4. Recent (last 6 months) history of regular menstrual cycles. Regular menstrual cycle meant the period of the cycle fell in the range of 21 to 35 days.
5. No contraceptive injection, implant, or intrauterine device within 6 months prior to the study and willing not to use any of them during the entire study period. Subject agreed to the use of a highly effective method of contraception throughout the study including:

   * 28-day regimens of combined oral contraceptives, patches, or rings
   * Bilateral tubal sterilization
   * Partner vasectomy
   * Condoms and spermicide
   * Diaphragm and spermicide At the discretion of the investigator, total abstinence was permitted as a method where age, lifestyle, or sexual orientation of the subject ensured compliance. If the subject was taking combined hormonal contraception, it had to be taken for at least 6 months prior to screening and be used throughout the duration of the study without interruption. No more than 50% of enrolled subjects were to be taking combined hormonal contraception.
6. Agreed not to use any dietary supplement or alternative medication intended to treat dysmenorrhea and/or its accompanying symptoms during the entire study period.
7. Was able to tolerate ibuprofen and willing to use only ibuprofen supplied by the sponsor for this study as a rescue medication.
8. Was able to understand and follow the study instructions, to complete the electronic subject diary, and to communicate with the investigator and staff.

Exclusion Criteria:

1. Known or suspected to have secondary dysmenorrhea due to pelvic inflammation, endometriosis, uterine myomata, ovarian pathological changes, or other pelvic diseases.
2. Known or suspected to have gastrointestinal or urological conditions that may cause abdominal/pelvic pain, such as colitis, appendicitis, irritable bowel syndrome, cholelithiasis, interstitial cystitis, urocystitis, nephrolithiasis, and other conditions that, according to the investigator's judgment, are not suitable for the study.
3. Use of an intrauterine contraceptive device, contraception injection, contraceptive implant, progesterone-only contraceptive pills, or an extended-cycle combined hormonal contraceptive regimen that does not foster cyclic withdrawal bleeding every 28 days within 6 months of screening or during the study.
4. Screening pelvic ultrasound findings suggestive of significant pathology including secondary causes of dysmenorrhea such as more than 2 uterine fibroids >3 cm in diameter, or complex ovarian cysts. At the discretion of the investigator, simple ovarian cysts <3 cm in diameter or functional ovarian cysts that were deemed to not require follow-up were permitted.
5. Obesity: body mass index (BMI) >32 kg/m2.
6. Positive gonorrhea and/or chlamydia test or evidence of other active sexually transmitted disease that, in the investigator's opinion, would make the subject not suitable for the study.
7. Known allergy to the study drug, or hypersensitivity to any of the study drug ingredients, or known allergy or intolerance to one or more of the excipients: β cyclodextrin and lactose, and according to the investigator's judgment, the allergy/intolerance was so severe that the subject was not suitable for the study.
8. Presence of one or more than one of the following: cerebrovascular disease, cardiovascular disease, pulmonary embolism, coagulopathy, thrombophlebitis, optic neuritis, retinal vein thrombosis, liver tumor, kidney tumor, renal failure, hepatitis, or other serious primary diseases of hepatic, renal or hematopoietic systems and mental disorders that according to the investigator's judgment renders the subject unsuitable for the study; or any chronic disease(s) for which the subject had been taking long term medication, and according to the investigator's judgment was unsuitable for the study. The investigator may have contacted the medical monitor and/or sponsor with questions about whether a subject was suitable for the study.
9. Hypertension, defined as sitting blood pressure (BP) systolic >140 mm Hg or diastolic >90 mm Hg (repetition of the measurement of BP was permitted to confirm the subject's hypertension condition).
10. Pregnant or trying to conceive during the study. Recent delivery, abortion, or lactation within 3 menstrual cycles before the start of treatment.
11. Alcoholism or drug abuse within the last 6 months prior to the study.
12. Regular use of any concomitant medications that might have confounded efficacy and/or safety assessments including, but not limited to, the following: narcotic, non NSAID, or NSAID analgesics for the treatment of conditions other than dysmenorrhea, psychotropic drugs, antidepressants, sedative hypnotics, sedating antihistamines, muscle relaxants, or tranquilizers. Selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors were permitted for indications other than pain provided that the subject had been on a stable dose for at least 2 menstrual cycles before providing consent for this study and agreed to remain on a stable dose throughout the course of the study.
13. Simultaneous participation in another clinical study or use of any experimental drug or device, or being a subject in another clinical research program within 30 days prior to the screening visit.
14. Use of any dietary supplement or alternative medication intended to treat dysmenorrhea or its accompanying symptoms within 30 days prior to the screening visit.
15. Major surgery scheduled for the study period.
16. Known to have a positive human immunodeficiency virus test.
17. Abnormal Papanicolaou (PAP) test results, except atypical squamous cells of unknown significance with reflex human papillomavirus test negative.
18. Inability to follow study procedures for any reason, including the following examples: language comprehension, psychiatric illness, or inability to get to the study center.
19. Had a clinically significant deviation from normal in any of the screening tests or examinations.
20. Had the presence of all 3 of the following signs and symptoms during the 2 weeks prior to screening.

    * Reported that her usual urine color was grade 7 or above on the pictorial scale (provided in the GF-2011-001 Special Assessment Guide) and laboratory examination of the color of her urine at screening confirmed this
    * Reported that she usually had dry stools and had experienced constipation for at least 2 consecutive days
    * Was noted on the screening examination by the investigator to have a red tongue with a yellow coating (example photograph provided in the GF 2011 001 Special Assessment Guide)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Song, MD, Study Director — Jiangsu Kanion Pharmaceutical Co., Ltd
Locations (23):
- United States (23):
  - Women's Health Research, Phoenix, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Women's Health Care at Frost Street, San Diego, California
  - Coastal Connecticut Research, New London, Connecticut
  - Atlanta Women's Research Institute, Inc., Atlanta, Georgia
  - Women's Healthcare Associates dba Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Chicago Research Center, Inc., Chicago, Illinois
  - Genesis Clinical Research, Fall River, Massachusetts
  - ClinSite, Ann Arbor, Michigan
  - Montana Medical Research, Missoula, Montana
  - Lawrence OB GYN Associates, Lawrenceville, New Jersey
  - The Center for Women's Health and Wellness LLC, Plainsboro, New Jersey
  - Suffolk OB-GYN, Port Jefferson, New York
  - Lynhurst Clinical Research, Winston-Salem, North Carolina
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Dial Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Advances in Health, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Women's Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KYG0395 (High Dose Group): KYG0395: 3 KYG0395 capsules tid (morning, midday, and evening)
- KYG0395 (Lower Dose Group): KYG0395: 3 KYG0395 capsules 2 times a day (bid) (morning and evening) plus 3 capsules of placebo (midday)
Period: Overall Study
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Started | 92 | 94 | 94
Overall Study | 92 | 94 | 94
Completed | 61 | 51 | 66
Not Completed | 31 | 43 | 28
Not completed — Adverse Event | 5 | 4 | 1
Not completed — Lost to Follow-up | 8 | 13 | 6
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 14 | 16 | 18
Not completed — Exclusion Criteria met during study | 2 | 1 | 0
Not completed — sponsor decision | 1 | 6 | 2

BASELINE CHARACTERISTICS:
Population: The number in the Flow is PPS data, consisted of all treatment completers from the FAS data set without any major protocol deviations leading to bias or misinterpretation of efficacy results. The FAS included all randomized subjects who at least received one dose of study treatments and had one valid post-baseline assessment of VAS score.
Groups:
- Total: Total of all reporting groups
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo | Total
Number analyzed (Participants) | 81 | 77 | 80 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.28) | 26.8 (5.18) | 27.3 (4.55) | 27.3 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 77 | 80 | 238
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 13 | 38
  Not Hispanic or Latino | 67 | 66 | 67 | 200
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 17 | 19 | 30 | 66
  White | 59 | 52 | 46 | 157
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to the End of Treatment Period in Maximum Dysmenorrheic Pain VAS Score
Description: VAS is represented by a straight line with extreme limits: from "no pain" and an associated image of a happy face at the left endpoint to "unbearable pain" and an associated image of an unhappy face at the right endpoint. The left endpoint is the minimum pain score of zero while the right endpoint is the maximum pain score of 100.
  The dysmenorrheic pain (lower abdominal cramping pain) that usually occurs just before and/or during menstruation was measured in this study using a The Visual Analogue Scale (VAS). Pain was assessed during 9 menstrual cycles from the beginning of the screening to the end of follow-up.
Time Frame: Baseline and end of treatment (6 months)
Population: Full analysis set: all subjects who received at least one treatment dose and had one post-baseline assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
units on a scale | -19.8 (2.84) | -18.0 (3.07) | -14.4 (2.86)
Statistical Analysis 1: Comparison: KYG0395 (High Dose Group) vs KYG0395 (Lower Dose Group) vs Placebo; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — p value for multiple comparison among 3 arms and comparison between investigational drug and placebo

2. Primary Outcome: The Change From Baseline in Number of Days With Dysmenorrheic Pain at the End of Treatment
Description: The change from baseline in number of days with dysmenorrheic pain at the end of 3 treatment cycles
Time Frame: Baseline and end of treatment (6 months)
Population: Full analysis set: all randomized subjects who received at least 1 dose of study treatments, and had at least 1 valid postbaseline assessment of dysmenorrheic pain VAS score
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
days | -1.4 (0.17) | -1.3 (0.19) | -1.1 (0.18)
Statistical Analysis 1: Comparison: KYG0395 (High Dose Group) vs KYG0395 (Lower Dose Group) vs Placebo; p value for multiple comparison among 3 arms and comparison between investigational drug and placebo; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

3. Primary Outcome: The Change From Baseline to the End of Follow-up Period in the Maximum VAS Score
Description: as for outcome 1
Time Frame: Baseline and end of follow-up (9 months)
Population: FAS: all randomized subjects who received at least 1 dose of study treatments, and had at least 1 valid postbaseline assessment of dysmenorrheic pain VAS score
Measure: Least Squares Mean (Standard Error); unit: unit of a scale
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
unit of a scale | -22.8 (2.93) | -15.5 (3.21) | -9.8 (2.79)
Statistical Analysis 1: Comparison: KYG0395 (High Dose Group) vs KYG0395 (Lower Dose Group) vs Placebo; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — p value for comparison between overall drug group vs placebo, and between high dose vs placebo

4. Primary Outcome: The Number of Days of Dysmenorrheic Pain at the End of Follow-up Period Compared With Baseline
Description: The change from baseline in the number of days with dysmenorrheic pain at the end of a 3-cycle follow-up period
Time Frame: Baseline and end of follow-up (9 months)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
days | -1.3 (0.19) | -1.5 (0.21) | -1.0 (0.18)
Statistical Analysis 1: Comparison: KYG0395 (High Dose Group) vs KYG0395 (Lower Dose Group) vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — p value for comparison between overall drug group vs placebo, and between low dose vs placebo

5. Secondary Outcome: Average Daily Dysmenorrheic Pain VAS Score at the End of Treatment and Follow-up Period
Description: as for outcome 1
Time Frame: Baseline, end of treatment (6 months) and end of follow-up (9 months)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
pills
  at the end of treatment | -14.7 (2.12) | -11.1 (2.29) | -9.6 (2.11)
  at the end of follow-up | -12.8 (2.15) | -10.1 (2.33) | -9.1 (2.04)

6. Secondary Outcome: Rescue Medication Consumption at the End of Treatment and Follow-up Period
Description: The change from baseline to the end of treatment and follow-up period in rescue medication consumption
Time Frame: Baseline, end of treatment (6 months) and end of follow-up (9 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 81 | 77 | 80
pills
  end of treatment | -2.6 (4.28) | -2.0 (4.1) | -2.0 (4.05)
  end of follow-up | -2.2 (4.66) | -2.6 (3.16) | -2.9 (3.93)

7. Secondary Outcome: Subject's Overall Satisfaction at the End of the 3-cycle Follow-up Period
Description: The subject's evaluation of overall satisfaction was recorded in the electronic subject diary at the end of the 3 treatment cycles and at the end of the 3-cycle follow-up period (at the end of the day before the subject goes to bed) using the numeric rating scale provided below:
  0=None, Not satisfied with the treatment outcome；
  1. Mild, Mildly satisfied with the treatment outcome；
  2. Most, Mostly satisfied with the treatment outcome；
  3. Complete, Completely satisfied with the treatment outcome.
Time Frame: Base line and end of follow-up (9 months)
Population: Full analysis set
Measure: Number; unit: percentage of complete satisfaction
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Number analyzed (Participants) | 59 | 49 | 62
percentage of complete satisfaction
  complete satisfaction | 35.6 | 16.3 | 24.2
  moderate satisfaction | 25.4 | 49.0 | 40.3
  mild satisfaction | 18.6 | 26.5 | 19.4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | KYG0395 (High Dose Group) | KYG0395 (Lower Dose Group) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/88 | 1/90 | 1/91
Other Adverse Events (participants affected / at risk) | 23/88 | 25/90 | 35/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KYG0395 (High Dose Group) (N=88) | KYG0395 (Lower Dose Group) (N=90) | Placebo (N=91)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Considered not related to study drug
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — considered not related to study drug as SAE occurred 30 days after the last study drug dose.
Abortion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — considered not related to study drug as SAE occurred 30 days after the last study drug dose.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KYG0395 (High Dose Group) (N=88) | KYG0395 (Lower Dose Group) (N=90) | Placebo (N=91)
any TEAE (Investigations) | 23 (23) | 23 (23) | 32 (32)
Gastrointestinal disorders (Gastrointestinal disorders) | 10 (10) | 9 (9) | 9 (9)
Infections and infestations (Infections and infestations) | 7 (7) | 7 (7) | 9 (9)
General disorders and administration site conditions (General disorders) | 1 (1) | 3 (3) | 6 (6)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Nervous system disorders (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other